CLINICAL TRIAL: NCT05091879
Title: Implementation and Evaluation of Preemptive Pharmacogenomics Testing in an Aging Population
Brief Title: Preemptive Pharmacogenomics Testing Among Geriatric Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2020-1103
Record Dates: First submitted 2021-09-27; First posted 2021-10-25 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Polypharmacy; Pharmacogenomic Testing
Keywords: pharmacogenomics; pharmacogenetics; Medicare; geriatric; multigene; polypharmacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): A multigene pharmacogenomics test will not be ordered for patients in this study arm, as is the standard of care.
- Pharmacogenomics Testing (Experimental): Patients in the experimental arm will be ordered a multigene pharmacogenomics test. This DNA test requires a blood draw, with the results expected to be reported in the medical record approximately 7 to 14 calendar days after the blood draw. These results will be made available to Geisinger healthcare professionals that have a treatment relationship with study participants.
  Interventions: Genetic: Multigene pharmacogenomics test

INTERVENTIONS:
Genetic: Multigene pharmacogenomics test — This multigene pharmacogenomics test will report genetic variation for genes that have Clinical Pharmacogenetics Implementation Consortium (CPIC) guidelines.
  Arms: Pharmacogenomics Testing

SUMMARY:
The primary goal of this study is to conduct pharmacogenomics testing (a type of DNA test) within an aging population and measure the impact of this test on medication selection, dosing, healthcare utilization, and costs of care.

DETAILED DESCRIPTION:
Pharmacogenomics is the study of how a patient's unique DNA may interact with medications that the patient currently takes or may take in the future. DNA may change how a patient reacts to a medication, such as changing how well it works or the side effects. Knowing a patient's DNA profile may help healthcare professionals select the best medication treatment plan to use. This could include selecting the best medication to give or the medication strength that will work best for the patient. Currently, there is no standard that helps healthcare professionals decide to order a pharmacogenomics test that includes multiple genes. The investigators of this study think that having these DNA results in the medical record for participants who are at least 65 years old and are taking 5 or more medications will result in better health since healthcare professionals may use these results for treatment planning. Knowing if this is true will help healthcare professionals decide if ordering this test will improve patient health.

This study seeks to recruit participants for a pharmacogenomic study who visit at Geisinger 65 Forward locations. Patients who meet the study requirements and consent to be enrolled in this study will be randomly put into a group that receives this pharmacogenomics test or a group that does not receive it. There is a 50% chance of being put in the group that receives this pharmacogenomics test. The investigators will follow all patients enrolled in this study as they visit with their healthcare providers in the future. Geisinger healthcare professionals will have access to the results of this test in the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Follows at a Geisinger 65 Forward clinic location
* Active prescriptions for 5 or more medications

Exclusion Criteria:

* Liver transplantation
* Allogenic hematopoetic stem cell transplantation
* Previously enrolled in the Electronic Medical Records and Genomics (eMERGE) pharmacogenomics cohort

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of pharmacogenomic results returned in patients' health records | Date of blood draw to test results reported in medical record, up to 1 month
  The primary objective will be assessed by comparing the total number of patients with returned results in the electronic health record (EHR) with the total number of tested patients.

SECONDARY OUTCOMES:
Composite of changes to medication therapy | Date of test results reported to end of study, up to 5 years
  The number of medication changes (e.g. dose or agent change) that healthcare professionals initiate due to pharmacogenomics return of results.
Number of hospitalizations | Date of test results reported to end of study, up to 5 years
  The number of hospitalizations patients encounter after receiving pharmacogenomics results
Number of ambulatory visits | Date of test results reported to end of study, up to 5 years
  The number of outpatient clinic visits patients encounter.
Costs of clinical care | Date of test results reported to end of study, up to 5 years
  The total healthcare costs of patients.
Medical costs of care | Date of test results reported to end of study, up to 5 years
  Measure of the costs of medical care (e.g. hospitalizations, outpatient visits, etc.), excluding pharmacy services.
Pharmacy costs of care | Date of test results reported to end of study, up to 5 years
  Measure of the costs of all pharmacy services (e.g. medications, consults, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Ryley Uber, Pharm.D., Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

REFERENCES:
- [Background] Mehta D, Uber R, Ingle T, Li C, Liu Z, Thakkar S, Ning B, Wu L, Yang J, Harris S, Zhou G, Xu J, Tong W, Lesko L, Fang H. Study of pharmacogenomic information in FDA-approved drug labeling to facilitate application of precision medicine. Drug Discov Today. 2020 May;25(5):813-820. doi: 10.1016/j.drudis.2020.01.023. Epub 2020 Feb 4. PMID 32032705
- [Background] Hicks JK, Bishop JR, Sangkuhl K, Muller DJ, Ji Y, Leckband SG, Leeder JS, Graham RL, Chiulli DL, LLerena A, Skaar TC, Scott SA, Stingl JC, Klein TE, Caudle KE, Gaedigk A; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for CYP2D6 and CYP2C19 Genotypes and Dosing of Selective Serotonin Reuptake Inhibitors. Clin Pharmacol Ther. 2015 Aug;98(2):127-34. doi: 10.1002/cpt.147. Epub 2015 Jun 29. PMID 25974703
- [Background] Hicks JK, Sangkuhl K, Swen JJ, Ellingrod VL, Muller DJ, Shimoda K, Bishop JR, Kharasch ED, Skaar TC, Gaedigk A, Dunnenberger HM, Klein TE, Caudle KE, Stingl JC. Clinical pharmacogenetics implementation consortium guideline (CPIC) for CYP2D6 and CYP2C19 genotypes and dosing of tricyclic antidepressants: 2016 update. Clin Pharmacol Ther. 2017 Jul;102(1):37-44. doi: 10.1002/cpt.597. Epub 2017 Feb 13. PMID 27997040
- [Background] Scott SA, Sangkuhl K, Stein CM, Hulot JS, Mega JL, Roden DM, Klein TE, Sabatine MS, Johnson JA, Shuldiner AR; Clinical Pharmacogenetics Implementation Consortium. Clinical Pharmacogenetics Implementation Consortium guidelines for CYP2C19 genotype and clopidogrel therapy: 2013 update. Clin Pharmacol Ther. 2013 Sep;94(3):317-23. doi: 10.1038/clpt.2013.105. Epub 2013 May 22. PMID 23698643
- [Background] Ramsey LB, Johnson SG, Caudle KE, Haidar CE, Voora D, Wilke RA, Maxwell WD, McLeod HL, Krauss RM, Roden DM, Feng Q, Cooper-DeHoff RM, Gong L, Klein TE, Wadelius M, Niemi M. The clinical pharmacogenetics implementation consortium guideline for SLCO1B1 and simvastatin-induced myopathy: 2014 update. Clin Pharmacol Ther. 2014 Oct;96(4):423-8. doi: 10.1038/clpt.2014.125. Epub 2014 Jun 11. PMID 24918167
- [Background] Dong OM, Wheeler SB, Cruden G, Lee CR, Voora D, Dusetzina SB, Wiltshire T. Cost-Effectiveness of Multigene Pharmacogenetic Testing in Patients With Acute Coronary Syndrome After Percutaneous Coronary Intervention. Value Health. 2020 Jan;23(1):61-73. doi: 10.1016/j.jval.2019.08.002. Epub 2019 Sep 25. PMID 31952675
- [Background] Ellenbogen MI, Wang P, Overton HN, Fahim C, Park A, Bruhn WE, Carnahan JL, Linsky AM, Balogun SA, Makary MA. Frequency and Predictors of Polypharmacy in US Medicare Patients: A Cross-Sectional Analysis at the Patient and Physician Levels. Drugs Aging. 2020 Jan;37(1):57-65. doi: 10.1007/s40266-019-00726-0. PMID 31782129
- [Background] Yang Y, Botton MR, Scott ER, Scott SA. Sequencing the CYP2D6 gene: from variant allele discovery to clinical pharmacogenetic testing. Pharmacogenomics. 2017 May;18(7):673-685. doi: 10.2217/pgs-2017-0033. Epub 2017 May 4. PMID 28470112
- [Background] Rohrer Vitek CR, Abul-Husn NS, Connolly JJ, Hartzler AL, Kitchner T, Peterson JF, Rasmussen LV, Smith ME, Stallings S, Williams MS, Wolf WA, Prows CA. Healthcare provider education to support integration of pharmacogenomics in practice: the eMERGE Network experience. Pharmacogenomics. 2017 Jul;18(10):1013-1025. doi: 10.2217/pgs-2017-0038. Epub 2017 Jun 22. PMID 28639489
- [Background] Bain KT, Schwartz EJ, Knowlton OV, Knowlton CH, Turgeon J. Implementation of a pharmacist-led pharmacogenomics service for the Program of All-Inclusive Care for the Elderly (PHARM-GENOME-PACE). J Am Pharm Assoc (2003). 2018 May-Jun;58(3):281-289.e1. doi: 10.1016/j.japh.2018.02.011. Epub 2018 Mar 27. PMID 29602745
- [Background] O'Donnell PH, Bush A, Spitz J, Danahey K, Saner D, Das S, Cox NJ, Ratain MJ. The 1200 patients project: creating a new medical model system for clinical implementation of pharmacogenomics. Clin Pharmacol Ther. 2012 Oct;92(4):446-9. doi: 10.1038/clpt.2012.117. Epub 2012 Aug 29. PMID 22929923
- [Background] Bain KT, Matos A, Knowlton CH, McGain D. Genetic variants and interactions from a pharmacist-led pharmacogenomics service for PACE. Pharmacogenomics. 2019 Jul;20(10):709-718. doi: 10.2217/pgs-2019-0047. Epub 2019 Aug 1. PMID 31368837
- See also: Clinical Pharmacogenetic Implementation Consortium (CPIC) guidelines. — https://cpicpgx.org/guidelines/
- See also: FDA Center for Drug Evaluation and Research Table of pharmacogenomic biomarkers in drug labeling. — https://www.fda.gov/drugs/science-and-research-drugs/table-pharmacogenomic-biomarkers-drug-labeling